## Statistical Analysis Plan (SAP) for the study

## Amino Acid Transport Imaging of Parathyroid Adenomas with anti-3-[18F] FACBC

Principal Investigator: David M Schuster, M.D.

IRB00051415

NCT01574287

Date: 06/13/2019

Data obtained from image ([18F]fluciclovine PET/CT and [99mTc]Sestamibi Planar (Early and Delayed) and Delayed SPECT/CT) interpretation were analyzed using SPSS version 23 (IBM, Armonk, NY).

Histopathologic confirmation of resected parathyroid adenoma or hyperplasia was reference standard for truth. Descriptive analysis was carried out, and mean  $\pm$  SD was reported as appropriate. Difference in means of uptake parameters for [18F]fluciclovine PET compared with [99mTc]sestamibi was determined using t-test. Statistical significance was set at p < 0.05.